CLINICAL TRIAL: NCT03116802
Title: Using Systems Vaccinology to Elucidate the Effects of Anti-inflammatory Therapy on Immune Response After Vaccination With a Live Attenuated Vaccine
Brief Title: Yellow Fever Vaccine on Statin/ Non Statin Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: YF-Statin-01
Record Dates: First submitted 2017-03-13; First posted 2017-04-17 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Yellow Fever Vaccine; Yellow Fever
MeSH Terms: conditions — Yellow Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Statin Group (Experimental): A total of 35 healthy adult subjects, 30-50 years old with a range of BMI from 18 to 30 kg/m2, pre-screened to be receiving long term statin therapy of ≥ 6 months and negative for diabetes (defined as HbA1c <6.5%) will be enrolled upon written informed consent. They will receive a single dose of 0.5ml of Stamaril (live attenuated yellow fever vaccine)
  Interventions: Drug: Stamaril (live attenuated yellow fever vaccine)
- Control Group (Active Comparator): Another 35 healthy non-diabetic adult subjects, 30-50 years old with a range of BMI from 18 to 30 kg/m2, not receiving long-term statins will serve as controls will be enrolled upon written informed consent.
  They will receive a single dose of 0.5ml of Stamaril (live attenuated yellow fever vaccine)
  Interventions: Drug: Stamaril (live attenuated yellow fever vaccine)

INTERVENTIONS:
Drug: Stamaril (live attenuated yellow fever vaccine) — They will receive a single dose of 0.5ml of Stamaril (live attenuated yellow fever vaccine)

SUMMARY:
Since the 1st pandemic of the 21st century caused by SARS coronavirus, the world has experienced outbreaks of swine origin H1N1 influenza, Ebola and Zika viruses, which have all resulted in global health crises. Rapid mass vaccination with an effective vaccine such as a live attenuated vaccine, of vulnerable immune-naïve populations to establish herd immunity is an approach to control outbreaks. Such live attenuated vaccine had been used with great success in sporadic yellow fever outbreaks and recently successfully employed in Ebola field trial, both of these diseases have the potential for pandemic spread. Indeed, live attenuated vaccines have proven especially effective in controlling childhood diseases and have even succeeded in eradicating polio and measles from most parts of the world. However, deployment of such vaccines for pandemic control cannot be limited to children but must include adults in order to rapidly elevate herd immunity rates to halt transmission. Vaccinating adults may produce efficacy rates significantly different to those observed in children due to the prevalence of chronic diseases and their associated metabolic complications. Presently, there are 1 billion people who are overweight, many suffer from concurrent metabolic disorders. As activation of the adaptive immunity is reliant on a robust innate immune response to vaccines, metabolic disorders and long-term anti-inflammatory therapy with interventions such as statins may reduce vaccine immunogenicity resulting in suboptimal efficacy in this subpopulation. This study would therefore test the hypothesis that statins reduce live attenuated vaccine immunogenicity. We will combine a clinical trial with systems vaccinology approaches to define the impact statins has on the innate immune, B and T-cell responses to live attenuated vaccination. Our study will thus extend upon another recently completed trial by us and will provide new insights into the determinants of vaccine efficacy in a rapidly growing and aging population globally

DETAILED DESCRIPTION:
Despite successful control of many infectious diseases since the 19th century, viral diseases remain an important and significant health burden in the 21st century. In fact, the turn of the 21st century saw the emergence of not only new but also re-emergent pathogens such as SARS, MERS, West Nile, Ebola, dengue and Zika viruses. In addition, the modern world is highly mobile and interconnected. The spread of infectious diseases is imminently only a flight away. It is thus of no surprise that epidemics in this century are happening at a much faster pace and spreading quicker to cause disruption to human health, society and the economy. Vaccination, particularly with a live attenuated vaccine (LAV), which has the most successful track record among the various forms of vaccines, remains the most economical public health tool available to prevent or stop the spread of infections and alleviate human sufferings. Rapid mass vaccination of at risk populations to establish herd immunity has been successfully employed to control sporadic YF outbreaks in Africa and South America. More recently, a clinical trial showed that ring vaccination of contacts with Ebola patients completely abrogated secondary virus spread. Vaccination in times of pandemics, however, cannot be limited to children but must include adults in order to rapidly elevate herd immunity rates to halt further transmission.

The use of LAV in adults has several important challenges that have not been systematically addressed. The population demographics in Singapore, like most developed countries have changed drastically over the past 3 decades. Along with improved nutrition, populations are now living longer but with increasing prevalence of chronic diseases such as obesity and dyslipidemia. Consequently, the anti-cholesterol group of drugs, with pleiotropic properties, statins, are among the commonest drugs prescribed globally for the prevention of secondary cardiovascular and major vascular complications. There is presently a mounting concern that the anti-inflammatory and immune-modulatory effects of statins could have a detrimental effect on vaccine efficacy. Indeed, studies examining inactivated influenza vaccination in older individuals had observed lower immunogenicity and overall efficacy with statin use. Whether statins have a similar negative immunogenicity effect on LAV remains undefined. The anti-inflammatory effects may dampen innate immune responses critical for triggering adaptive immunity resulting in reduced immunogenicity. Conversely, the suppression of innate immune responses could favor LAV infection and replication, allowing adaptive immune cells a longer period to sense the antigen, become activated and differentiated for improved immune response.

In this study, an experimental medicine investigation that leverages on a recently completed clinical trial that the PI led examining how cross-reactive antibodies altered the immunogenicity of yellow fever (YF) vaccination. We will seek to clarify the effects of statin on LAV immunogenicity. YF vaccine is an excellent LAV, which remains the WHO recommended response to the ever-present threat of YF outbreak. It has also served as an important model for studying human antiviral immunity. We propose to test the hypothesis that long term statins therapy alters YF LAV immunogenicity by coupling the power of a clinical trial with comprehensive systems vaccinology to define the impact statins have on the adaptive immune response to YF vaccination. This study will elucidate how statins modulate the networks that drive immunity to vaccination in a fast growing population globally. Knowledge on how statins impact LAV immunogenicity would inform public health authorities on the size of the general population that should be vaccinated to compensate for alterations in immunogenicity in this subpopulation to achieve sufficient herd immunity for epidemic and pandemic control.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 30-50 years of age at the time of screening.
2. Negative for diabetes (defined as HbA1c <6.5%)
3. Range of BMI from 18 to 30kg/m 2
4. Statin Group: receiving long term statin therapy (Simvastatin, Atorvastatin and Rosuvastatin) for ≥6 months
5. Control group: not receiving long-term statins
6. Negative for anti-dengue antibodies by ELISA. Subjects will be screened using a commercially available ELISA (PanBio)
7. Subjects who are willing to comply with the requirements of the study protocol and scheduled visits. (e.g., completion of the subject diary, return for follow-up visits) and who are willing to make themselves available for the duration of the study, with access to a consistent means of telephone contact, which may be either at home or at the workplace, land line, or mobile, but NOT a pay phone or other multiple-user device (i.e. a common-use phone serving multiple rooms or apartments).
8. Subjects who give written informed consent approved by the Ethical Review Board governing the site.
9. Satisfactory baseline medical assessment as assessed by physical examination and a stable health status. The laboratory values must be within the normal range of the assessing site or show abnormalities that are deemed not clinically significant as judged by the investigator. A stable health status is defined as the absence of a health event satisfying the definition of a serious adverse event.
10. Accessible vein at the forearm for blood collection.
11. Female subjects of non-child bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause. Post menopause: subjects must have had at least 12 months of natural (spontaneous) amenorrhea
12. Female subjects of childbearing potential may be enrolled in the study if they have negative urine pregnancy tests on the day of screening and day of vaccination
13. Both male (if he has a partner of childbearing potential) and female subjects (of childbearing potential) must agree to use adequate and reliable contraceptive measures (eg. Spermicides, condoms, contraceptive pills) or practice abstinence for 10 days after vaccination

Exclusion Criteria:

1. Presence of acute infection in the preceding 7 days or presence of a temperature ≥ 38.0°C (oral or tympanic temperature assessment), or acute symptoms greater than of "mild" severity on the scheduled date of first vaccination.
2. History of severe drug and /or food allergies and/or known allergies to the trial product or its components.
3. Any condition that, in the opinion of the investigator, would complicate or compromise the study or wellbeing of the subject.
4. Woman who is pregnant or breast feeding.
5. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, neuropsychiatric, or immunosuppressive disorders that would be a risk factor when administered the Investigational product (IP).
6. History of thymus gland disease.
7. Diagnosed with cancer or on treatment for cancer within the 3 years prior to the screening.
8. Evidence of clinically significant anaemia and other any significant active haematological disease, or having donated > 450 mL of blood within the past three months.
9. Evidence of substance abuse, or previous substance abuse.
10. Participation in a study involving administration of an investigational compound within the past four months, or planned participation during the duration of this study.
11. Administration of any licensed vaccine within 30 days before the first study vaccine dose.
12. Subject who has been vaccinated with YF vaccine previously.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
the adaptive immune response to YF vaccination in (A): Adult human volunteers who are on long term statins therapy and (B): Adult human volunteers (controls) | 28 days
  the difference in neutralizing antibody titer to YF17D at Day 28, as measured by plaque reduction neutralization test (PRNT)

SECONDARY OUTCOMES:
the difference in innate immune response to YF vaccination in adult human volunteers on long term statins therapy compared to controls post-YF vaccination | 28 days
  viremia levels response in adult human volunteers on long term statins therapy compared to controls post-YF vaccination
the cellular immune response of adult human volunteers on long term statins therapy with controls following YF vaccination. | 28 days
  To examine the Cd4+ and Cd8+ T cell response in adult human volunteers on long term statins therapy compared to controls post-YF vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Dr Low, Principal Investigator — Singapore General Hospital
Locations (1):
- SingHealth Investigational Medicine Unit, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No